CLINICAL TRIAL: NCT05220852
Title: Effects of Dry Needling With a Standard Exercise Programme on Pain and Quality of Life in Patients With Chronic Mechanical Neck Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Muhannad Abdulrahman Almushahhim, Principal Investigato, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-PGS-2021-03-209
Record Dates: First submitted 2021-12-03; First posted 2022-02-02 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain | interventions — Dry Needling; Exercise

STUDY DESIGN:
Intervention Model Description: RTC single-blind
Who Masked: Participant
Masking Description: all the research subjects were masked and enrolled by picking up one of two sealed envelope to take place in one of the groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling and exercise (Experimental): Subjects in this group will undergo one session of dry needling in their upper trapezius muscles to address any overactive trigger points, and they will subsequently continue with neck exercises for a minimum of two weeks, three times per week.
  Interventions: Combination Product: Dry needling with exercise
- Exercise (Active Comparator): subjects in this group will have neck exercise only for 2 weeks minimum 3 times a week.
  Interventions: Other: Exercise

INTERVENTIONS:
Combination Product: Dry needling with exercise — At the initial session, dry needling will be given to their upper trapezius muscles' hyperactive trigger sites, and EX will continue for a minimum of three times per week.
  1. Cranio-cervical spine flexion is the exercise.
  2. Extension of the cranio-cervical spine Exercice 3 Shoulder Elevation 4-Retraining of the scapular muscles Every exercise should be done for 30 se
  Arms: Dry needling and exercise
Other: Exercise — patients in this group are going to have onley neck exercise for 2 weeks minimum 3 times a week.
  1. Cranio-cervical spine flexion is the exercise.
  2. Extension of the cranio-cervical spine Exercice 3 Shoulder Elevation 4-Retraining of the scapular muscles Every exercise should be done for 30 se
  Arms: Exercise

SUMMARY:
Abstract\sBackground

Physical therapists frequently utilize dry needling (DN), which focuses on trigger points and non-trigger point structures, to treat mechanical neck pain (MNP). It is an invasive procedure that involves inserting solid fiber needles into myofascial trigger points or hyperirritable nodules that are painful to the touch. This procedure can affect the motor and autonomic neurons and relieve pain.

Objectives

examining the short-term effects of dry needling in combination with a standardized exercise program on pain and quality of life in chronic mechanical neck pain

Methods

The allocation of 18 participants to the DN or Exercise intervention groups will be done at random. Before the exam, the Beck Depression Inventory (BDI), Neck Disability Index (NDI), Short Form-36 Quality of Life Scale, and Numerical Rating Scale (NPS-11) will be evaluated.

Analytical Statistics

For the statistical analysis of the data, SPSS 23.0 will be employed. The "Kolmogorov-Smirnov test" will be used to determine whether the data are distributed normally. The effectiveness of each intervention will be determined using a paired t test, and between-group comparisons will be made using an independent t test. The distribution of categorical variables will be compared using a chi-square test. A 95% confidence interval and p0.05 will be used to determine significance.

Key words: mechanical neck pain, dry needling, neck exercises, and quality of life.

DETAILED DESCRIPTION:
Procedure

The lead investigator screened the participants to ensure that they met the requirements for participation in the study.

The participants were randomly divided into the "control group" and the "experimental group."

Intervention

Needling dry

The experimental group will receive dry needling in addition to the exercise routine, while the control group will just receive the exercise protocol.

The trigger point (TrP) DN will be used, and a TrP location will be palpated and designated for needle insertion in the upper trapezius muscle. Stainless-steel disposable needles 0.3 30 mm; Novasan, S.A.

The needle will be placed into the skin for up to 10 to 15 mm, until a local twitch reaction is felt, and the person will be monitored for two weeks after that. For two weeks, the participant will begin the workouts once daily.

Protocol for neck exercise:

Both the experimental and control groups will get a standardized workout regimen that included neck and upper back muscular stretching and strengthening.

Confidentiality:

Data will be collected collectively and maintained confidentially in a computer protected by a password; no individual's name will be revealed.

ELIGIBILITY:
Inclusion Criteria:

-Participants who have been given a primary care doctor's or an orthopaedic consultant's medical diagnosis of chronic mechanical neck discomfort will be screened by the lead investigator.

2- Participants who were diagnosed with chronic neck discomfort that was brought on by neck movements, postures, and cervical palpation 3. Neck ache that has persisted for longer than a month. 4- Participants must not be receiving any treatment for their persistent neck discomfort at the time they are recruited for the study.

Exclusion Criteria:

- Neurologic impairments are symptoms of radiculopathy, according to participants.

* Medical diagnosis of cervical myelopathy or radiculopathy

  . Aversion to needles
* A history of shoulder, whiplash, or cervical spine injuries that was reported. Any "red flags" (malignancy, inflammatory arthritis, fracture, osteoporosis, and others).

patient with a congenital condition

- Any treatment that research participants may have been receiving at the time of recruitment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — 18-60
Enrollment: 31 (Actual)
Dates: Start 2022-02-06 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-08-09 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale | 2 times From admission to discharge, up to 2 week (pre first intervention and post last intervention)
  used to assess the intensity of the pain , the NPS ranges between 0 and 10 (0: minimum pain, 10: maximum pain).
"Short Form-36 Quality of Life Scale (SF-36 QOLS) | 2 times From admission to discharge, up to 2 week (pre first intervention and post last intervention)
  for assessing the physical functions of the body through analysis of body pain, physical role difficulties (PRD), vitality/energy, the general perception of health, social functions and mental health. The sub-scores will be calculated separately between 0 and 100 (0: the worst, 100: the best health status)
Beck Depression Inventory (BDI) | 2 times From admission to discharge, up to 2 week (pre first intervention and post last intervention)
  To assess patient depression,The total score of BDI were evaluated between 0 and 63. BDI scores near to high range or above than that indicate more severe forms of depression
The functional disability, Neck Disability Index (NDI) | 2 times From admission to discharge, up to 2 week (pre first intervention and post last intervention)
  has been designed to assess the pain intensity of the neck and how it affects the quality of life by affecting daily activities. The total NDI score is 0 and 54 and consists of 10 questions.(less score less disability)

CONTACTS AND LOCATIONS:
Locations (1):
- Imam Abdulrahman Bin Faisal University, Dammam, Eastern Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Abbaszadeh-Amirdehi, M. et al. (2017) 'Therapeutic Effects of Dry Needling in Patients with Upper Trapezius Myofascial Trigger Points', Acupuncture in Medicine, 35(2), pp. 85-92. doi: 10.1136/acupmed-2016-011082. 2. Alghadir, A. H., Anwer, S. and Iqbal, Z. A. (2016) 'The psychometric properties of an Arabic numeric pain rating scale for measuring osteoarthritis knee pain', Disability and Rehabilitation, 38(24), pp. 2392-2397. doi: 10.3109/09638288.2015.1129441. 3. Andersen, L. L. et al. (2011) 'Prevalence and anatomical location of muscle tenderness in adults with nonspecific neck/shoulder pain', BMC Musculoskeletal Disorders, 12(1), p. 169. doi: 10.1186/1471-2474-12-169. 4. 'ASAP_Guidelines_2013.pdf' (no date). Available at: https://www.dryneedling.com.au/wp-content/uploads/2016/01/ASAP_Guidelines_2013.pdf (Accessed: 28 March 2020). 5. Beck, A. T. et al. (1961) 'An inventory for measuring depression', Archives of General Psychiatry, 4, pp. 561-571. doi: 10.1001/archpsyc.1961.01710120031004. 6. Borg-Stein, J. (2004) 'Musculoskeletal head and neck pain', Seminars in Pain Medicine, 2(2), pp. 85-92. doi: 10.1016/j.spmd.2004.04.004. 7. Brady, S. et al. (2014) 'Adverse events following trigger point dry needling: a prospective survey of chartered physiotherapists', Journal of Manual & Manipulative Therapy, 22(3), pp. 134-140. doi: 10.1179/2042618613Y.0000000044. 8. Cerezo-Téllez, E. et al. (2016) 'Effectiveness of dry needling for chronic nonspecific neck pain: a randomized, single-blinded, clinical trial', PAIN, 157(9), pp. 1905-1917. doi: 10.1097/j.pain.0000000000000591. 9. Cross, K. M. et al. (2011) 'Thoracic Spine Thrust Manipulation Improves Pain, Range of Motion, and Self-Reported Function in Patients With Mechanical Neck Pain: A Systematic Review', Journal of Orthopaedic & Sports Physical Therapy, 41(9), pp. 633-642. doi: 10.2519/jospt.2011.3670. 10. Fawzi, M. H., Fawzi, M. M. and Abu-Hindi, W. (2012) 'Arabic version of the Major Depression Inventory as a diagnostic tool: reliability and concurrent and discriminant validity.', Eastern Mediterranean health journal = La revue de sante de la Mediterranee orientale = al-Majallah al-sihhiyah li-sharq al-mutawassit. doi: 10.26719/2012.18.4.304. 11. Geneen, L. J. et al. (2017) 'Physical activity and exercise for chronic pain in adults: an overview of Cochrane Reviews', The Cochrane Database of Systematic Reviews, 2017(4). doi: 10.1002/14651858.CD011279.pub3. 12. Gerber, L. H. et al. (2015) 'Dry Needling Alters Trigger Points in the Upper Trapezius Muscle and Reduces Pain in Subjects with Chronic Myofascial Pain', PM & R : the journal of injury, function, and rehabilitation, 7(7), pp. 711-718. doi: 10.1016/j.pmrj.2015.01.020. 13. Graham, N. et al. (2008) 'Mechanical traction for neck pain with or without radiculopathy', Cochrane Database of Systematic Reviews, (3). doi: 10.1002/14651858.CD006408.pub2. 14. Gross, A. et al. (2010) 'Manipulation or mobilisation for neck pain: A Cochrane Review', Manual Therapy, 15(4), pp. 315-333. doi: 10.1016/j.math.2010.04.002. 15. Gross, A. et al. (2015) 'Exercises for mechanical neck disorders', The Cochrane database of systematic reviews, 1, p. CD004250.